CLINICAL TRIAL: NCT03382210
Title: Impact of a Colorectal Enhanced Recovery Program Implementation on Clinical Outcomes and Institutional Costs: A Prospective Cohort Study With Retrospective Control
Brief Title: Impact of a Colorectal Enhanced Recovery Program Implementation on Clinical Outcomes and Institutional Costs
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Ministero della Salute, Italy (Other); Università degli Studi di Ferrara (Other)
Responsible Party: Sponsor
Other Study IDs: RF-2010-2322017
Record Dates: First submitted 2017-11-06; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Colorectal Surgery; Recovery of Function; Laparoscopic Surgery
Keywords: Enhanced Recovery Program

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERP group: A prospective series of patients (N=100) undergoing elective colorectal resection and completing a standardized enhanced recovery protocol in 2013-2015 (ERP group) at the S. Anna University Hospital in Ferrara (Italy).
  Interventions: Other: Enhanced recovery protocol
- Pre-ERP group: A retrospective series of patients (N=100) operated on at the the S. Anna University Hospital in Ferrara (Italy) in 2009-2011 (Pre-ERP group), before the introduction of ERP methodology.

INTERVENTIONS:
Other: Enhanced recovery protocol — Standardized enhanced recovery protocol including 21 perioperative items.
  Groups: ERP group

SUMMARY:
Importance: The Enhanced Recovery Program (ERP) for perioperative care of the surgical patient reduces the postoperative metabolic response and organ dysfunction thereby accelerating functional recovery. Consequently, the hospital length of stay (LOS) may be reduced, with no increase in morbidity and mortality rates resulting in a potential economic benefit.

Objective: To determine impact on postoperative recovery and cost-effectiveness of implementing an ERP for colorectal surgery in an Italian academic center.

Design, Setting, and Participants: A prospective consecutive series of patients (N=100) undergoing elective colorectal resection completing a standardized ERP in 2013-2015 (ERP group) will be compared to patients (N=100) operated on at the same Italian University hospital in 2010-2011 (Pre-ERP group) before introducing ERP program. The exclusion criteria are: age>80 years old, ASA score IV, tumour stage IV, and inflammatory bowel disease.

Exposures: ERP for perioperative care. Main Outcomes and Measures: To evaluate the impact of colorectal ERP implementation on hospital LOS proxy of functional recovery. Secondary outcomes include: postoperative complications, 30-day readmission and mortality, protocol adherence, nursing workload, cost-effectiveness, and factors predicting prolonged hospital LOS. Patients' satisfaction in ERP group will also be prospectively evaluated.

DETAILED DESCRIPTION:
Introduction The Enhanced Recovery Program (ERP) is a scientific evidence-based perioperative care approach based on multidisciplinary team working and multimodal methodology, with the aim to reduce metabolic response to surgical stress and organ dysfunction induced by surgery, thereby accelerating postoperative recovery. Consequently, the hospital length of stay (LOS) after surgery would be significantly reduced, with no increase in morbidity and mortality rates 2-4 resulting in a potential economic benefit.

Although the concept of enhancing recovery after surgery implementing specific pathways is now widely recognized, the diffusion of ERPs is still limited to Northwestern Europe, USA, and Canada, and slightly less common in Southern Europe, where it prevails in Spain, Portugal, and Italy.

The implementation of an ERP relies on the establishment of a motivated multidisciplinary team including surgeons, anesthesiologists, and nurses who agree on the end points of management and act in close coordination throughout the perioperative phases (outpatients clinic, preoperative unit, operating theater, postoperative recovery room, surgical ward). It has been shown that compliance to the elements of the ERP protocol correlates with clinical outcomes.

The aim of this study is three-fold: 1) to investigate the impact of the colorectal ERP implementation in an Italian University hospital, on postoperative recovery, evaluating the efficacy (functional recovery, LOS), the safety (postoperative complications, 30-day readmission and mortality), the adherence to the protocol, the nursing workload, and the cost-effectiveness; 2) to assess the predictive factors of prolonged hospital LOS after colorectal resection; and 3) to measure patients' satisfaction in the ERP group.

Methods A prospective series of patients (N=100) undergoing elective colorectal resection and completing a standardized ERP in 2013-2015 (ERP group) at the S. Anna University Hospital in Ferrara (Italy) will be compared to a retrospective series of patients (N=100) operated on at the same academic hospital in 2009-2011 (Pre-ERP group), and before the introduction of ERP methodology. The Italian Ministry of Health will fund this study, which will begin in January 2013. In 2012 the ERP multidisciplinary team was built, the ERP protocol was prepared, and informative meetings were scheduled. All consecutive patients between the ages of 18 and 79 years of age and scheduled for elective colorectal resection will be enrolled for the study. The exclusion criteria for both groups are: age >80 years old, American Society of Anesthesia (ASA) score IV, Tumour Node Metastasis (TNM) stage IV, inflammatory bowel disease.

The criteria adopted for discharge of the ERP group patients are the same applied to the Pre-ERP group patients, specifically: 1) unrestricted oral diet, 2) full intestinal function recovery (i.e. passage of flatus and stool), 3) dynamic pain control (Numerical Rate Scale ≤3) by oral analgesia, 4) independent walking, and 5) no signs of infection.

In order to evaluate the impact on postoperative recovery of the colorectal ERP implementation, the hospital LOS, a proxy of functional recovery, is adopted as a primary outcome. Secondary outcomes are postoperative complications, 30-day readmission and mortality, adherence to the protocol, nursing workload, cost-effectiveness, and the predictive factors of prolonged hospital LOS.

All the data for the study will be collected prospectively for the ERP group and retrospectively for the Pre-ERP group.

ERP group All patients will be extensively informed about the ERP, including discharge criteria and 4-day planned hospital LOS, by thorough preoperative counseling and an illustrated booklet specifically developed and validated by the multidisciplinary team will be explained and given to patients. Although laparoscopy will be preferred, the surgical approach will be discussed with the patient. A converted laparoscopy is defined as unplanned extension of the surgical incision.

All patients in the ERP group will be encouraged during hospitalization to follow the perioperative protocol, and they will be informed about the objectives to be achieved on each day of hospital stay, including the discharge home.

All ERP elements included in the colorectal protocol will be prospectively recorded and checked if successfully achieved (i.e., protocol compliance) by a detailed care program (daily care map) for each postoperative day (POD).

Pre-ERP group All patients were treated following traditional perioperative care principles based on: 1-2) preoperative fasting since midnight with no carbohydrate loaded drinks; 3) opioid-based anesthesia with or without thoracic epidural; 4) postoperative pain control with intravenous opioids and/or thoracic epidural and/or non-steroidal anti-inflammatory drugs (NSAIDs); 5-6) nasogastric tube (NGT) removal and oral feeding at restoration of intestinal activity; 7) abdominal drain removal at bowel movements; 8) mobilization at patient's will; and 9) bladder catheter removal at full mobilization.

Preoperative counseling focused on patient's training, daily goals assignment or predefined day of discharge were not planned.

The medical records will be reviewed to evaluate adherence to any of the elements comprised in the ERP protocol and to determine how much the clinical practice has been modified by its implementation.

Fulfillment of the predefined discharge criteria will be checked in both study groups, and outpatient appointment was scheduled at 15 and 30 days after the operation.

The nursing workload will be evaluated using the Project Recherche Nursing (PRN), a standardized and validated point system based on eight groups of activities (respiration, feeding and hydration, elimination, hygiene, mobilization, communication, treatments, diagnostic procedures) that was developed in Canada to measure the level of patients' nursing care required. The PRN value will be compared between groups for the first few days of hospital stay based on the ERP patients' median LOS, the higher the point value the greater the amount of direct care required.

To determine the costs-effectiveness of the ERP versus traditional care we will collect costs on: 1) ERP implementation; 2) preoperative phase (i.e. preoperative counseling, booklet); 3) direct cost of hospitalizations (i.e. operating room, drugs, exams, visits, LOS); 4) re-hospitalizations.

To evaluate the patients' satisfaction, Patient Satisfaction Consultation Questionnaire (PSCQ-7) and the Core Questionnaire Patient Satisfaction (COPS) will be administered to all ERP group patients at hospital discharge.

The study will be conducted in accordance with the principles of Helsinki Declaration, with approval of the medical ethics review board of the S. Anna University Hospital. A written informed consent will be obtained from all enrolled patients.

Statistical analysis Data will be expressed as median (InterQuartile Range 25-75) and mean±standard deviation according to distribution assessed by Shapiro-Wilk test. Categorical data will be presented as number. Data will be analyzed using Chi-square, t-student, and Mann-Whitney tests as appropriate. Kaplan-Meier method has been used for analysis of surgical operation duration and hospital LOS. Log-Rank test has been employed to compare duration of surgical operation, time to functional recovery, and hospital LOS between groups. We will assess the association of different baseline characteristics, intraoperative variable and type of perioperative protocol with prolonged hospital LOS in the univariate Cox regression analysis adopting time to patients' hospital discharge as the endpoint of interest. For the time to event analyses, patients will be censored at time of hospital discharge. We will then calculate multivariate Cox regression analyses adjusted for potential confounders to assess independent predictors of prolonged hospital LOS. Of note, hazard ratios (HRs) <1 will correspond to an association of the factor with prolonged hospital LOS, while HRs >1 correspond to earlier discharge. Significance will be considered for values of p <0.05. Statistical analysis will performed with IBM Statistics for Windows (IBM Corp.).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective colorectal resection at the S. Anna University Hospital in Ferrara (Italy)

Exclusion Criteria:

* age >80 years old,
* American Society of Anesthesia (ASA) score IV,
* TNM stage IV,
* inflammatory bowel disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective colorectal resection at the S. Anna University Hospital in Ferrara (Italy) between 2013-2015 (ERP group) and 2009-2011 (Pre ERP group)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01-11 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2016-04-11 (Actual)

PRIMARY OUTCOMES:
Postoperative Hospital Length Of Stay (LOS). | Within 10 days from date of surgical operation.
  The postoperative hospital LOS, proxy of functional recovery, is defined as the number of days from the date of surgical operation to the date of hospital. Patients in both study groups wil be discharged from the hospital upon reaching all predefined discharged criteria. For the ERP group it is estimated a 4 to 5-day hospital LOS according to the protocol, while in the traditional group an 8 to 10-day hospital stay is expected.

SECONDARY OUTCOMES:
Morbidity. | Within 30 days from date of surgical operation.
  Postoperative complications.
Mortality. | Within 30 days from date of surgical operation.
  Postoperative mortality rate.
30-day readmission. | Within 30 days from date of surgical operation.
  30-day readmission rate to the hospital.
Nursing workload evaluated by Project de Recherche en Nursing (PRN). | From date of surgical operation to the 4th postoperative day.
  Nursing workload for postoperative patient care.
Cost-effectiveness. | From date of preoperative counseling to 30 days from date of surgical operation.
  Direct cost analysis.
Predictors of prolonged LOS. | Within 10 days from date of surgical operation.
  Assessment of the association of different baseline characteristics, intraoperative variable and type of perioperative protocol with prolonged hospital LOS in the univariate Cox regression analysis adopting time to patients' hospital discharge as the endpoint of interest. The hospital LOS is defined as the number of days from the date of surgical operation to the date of hospital discharge. Patients in both study groups wil be discharged from the hospital upon reaching all predefined discharged criteria. The estimated hospital LOS is 4 to 5 days in ERP group and 8 to 10 days in the traditional group.
ERP patients' satisfaction 1. | Within 40 days from date of preoperative counseling.
  Patients' satisfaction in ERP group will be assessed by the Patient Satisfaction Consultation Questionnaire (PSCQ-7). Due to the retrospective nature of the control group, the questionnaire wil be submitted only to ERP group patients on the day of hospital discharge and will evaluate patients' care since the date of preoperative counseling. Preoperative conseling occurs about 30 days before the surgical operation. The estimated hospital LOS is 4 to 5 days in ERP group and 8 to 10 days in the traditional group.
ERP patients' satisfaction 2. | Within 40 days from date of preoperative counseling.
  Patients' satisfaction in ERP group will be assessed by Core Questionnaire Patient Satisfaction (COPS). Due to the retrospective nature of the control group, the questionnaire wil be submitted only to ERP group patients on the day of hospital discharge and will evaluate patients' care since the date of preoperative counseling. Preoperative conseling occurs about 30 days before the surgical operation. The estimated hospital LOS is 4 to 5 days in ERP group and 8 to 10 days in the traditional group.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo V Feo, MD, Principal Investigator — University Hospital Ferrara

IPD SHARING:
Plan to Share IPD: Undecided
Formal requests will be individually evaluated

REFERENCES:
- [Background] Varadhan KK, Neal KR, Dejong CH, Fearon KC, Ljungqvist O, Lobo DN. The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery: a meta-analysis of randomized controlled trials. Clin Nutr. 2010 Aug;29(4):434-40. doi: 10.1016/j.clnu.2010.01.004. Epub 2010 Jan 29. PMID 20116145
- [Background] Greco M, Capretti G, Beretta L, Gemma M, Pecorelli N, Braga M. Enhanced recovery program in colorectal surgery: a meta-analysis of randomized controlled trials. World J Surg. 2014 Jun;38(6):1531-41. doi: 10.1007/s00268-013-2416-8. PMID 24368573
- [Background] Braga M, Pecorelli N, Scatizzi M, Borghi F, Missana G, Radrizzani D; PeriOperative Italian Society. Enhanced Recovery Program in High-Risk Patients Undergoing Colorectal Surgery: Results from the PeriOperative Italian Society Registry. World J Surg. 2017 Mar;41(3):860-867. doi: 10.1007/s00268-016-3766-9. PMID 27766398
- [Background] Adamina M, Kehlet H, Tomlinson GA, Senagore AJ, Delaney CP. Enhanced recovery pathways optimize health outcomes and resource utilization: a meta-analysis of randomized controlled trials in colorectal surgery. Surgery. 2011 Jun;149(6):830-40. doi: 10.1016/j.surg.2010.11.003. Epub 2011 Jan 14. PMID 21236454
- [Background] Lee L, Mata J, Ghitulescu GA, Boutros M, Charlebois P, Stein B, Liberman AS, Fried GM, Morin N, Carli F, Latimer E, Feldman LS. Cost-effectiveness of Enhanced Recovery Versus Conventional Perioperative Management for Colorectal Surgery. Ann Surg. 2015 Dec;262(6):1026-33. doi: 10.1097/SLA.0000000000001019. PMID 25371130
- [Background] Frostholm L, Fink P, Oernboel E, Christensen KS, Toft T, Olesen F, Weinman J. The uncertain consultation and patient satisfaction: the impact of patients' illness perceptions and a randomized controlled trial on the training of physicians' communication skills. Psychosom Med. 2005 Nov-Dec;67(6):897-905. doi: 10.1097/01.psy.0000188403.94327.5b. PMID 16314594
- [Background] Kleefstra SM, Kool RB, Veldkamp CM, Winters-van der Meer AC, Mens MA, Blijham GH, de Haes JC. A core questionnaire for the assessment of patient satisfaction in academic hospitals in The Netherlands: development and first results in a nationwide study. Qual Saf Health Care. 2010 Oct;19(5):e24. doi: 10.1136/qshc.2008.030825. Epub 2010 Jun 24. PMID 20577001
- [Background] Feo CV, Portinari M, Tsolaki E, Romagnoni G, Verri M, Camerani S, Volta CA, Mascoli F. The effect of an Enhanced Recovery Program in elective retroperitoneal abdominal aortic aneurysm repair. J Vasc Surg. 2016 Apr;63(4):888-94. doi: 10.1016/j.jvs.2015.09.060. Epub 2016 Jan 21. PMID 26806521
- [Result] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305